CLINICAL TRIAL: NCT06355596
Title: Development and Validation of a Virtual Teaching Method for Minimally Invasive Surgery Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 20IC6361
Record Dates: First submitted 2024-03-19; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Surgery
Keywords: Laparoscopic surgery skills; Medical education; Minimally invasive surgery

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated to either face-to-face or virtual teaching groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-face teaching (Active Comparator): Face-to-face teaching of laparoscopic skills
  Interventions: Other: Virtual teaching
- Virtual teaching (Experimental): Virtual teaching of laparoscopic skills
  Interventions: Other: Virtual teaching

INTERVENTIONS:
Other: Virtual teaching — Virtual teaching of laparoscopic skills

SUMMARY:
The goal of this observational study is to develop and evaluate a virtual teaching method for minimally invasive surgery (MIS) skills among novice learners, using widely available technology and incorporating objective assessments of proficiency. The main questions it aims to answer are:

Can MIS skills be effectively taught to novice learners through a virtual platform using widely available technology? How do virtual and face-to-face (F2F) teaching methods compare in terms of effectiveness, measured by performance in MIS tasks and cognitive workload parameters?

Participants in this study will:

Be randomly allocated to either F2F or virtual teaching groups. Undergo training and evaluation using validated laparoscopic assessments, namely the McGill Inanimate System for Training and Evaluation of Laparoscopic Skills (MISTELS) peg transfer task and the European Academy laparoscopic 'Suturing Training and Testing' (SUTT) assessment.

Have their performance and cognitive workload parameters (SURG-TLX score, heart rate, and pupil metrics) evaluated during the tasks.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age > 18)
* Medical student, Foundation Year or Core Trainee level or equivalent

Exclusion Criteria:

* Specialty Registrar level
* Consultant level

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
McGill Inanimate System for Training and Evaluation of Laparoscopic Skills (MISTELS) peg transfer task score | Two days
  Time to completion of task (minutes)
European Academy laparoscopic 'Suturing Training and Testing' (SUTT) assessment score | Two days
  Time to completion of task (minutes)

SECONDARY OUTCOMES:
SURG-TLX score | Two days
  Workload score ranging from 0 to 100
Heart rate | Two days
  Beats per minute
Pupil metrics | Two days
  Mean pupil size (mm) and blinks per minute

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No